CLINICAL TRIAL: NCT02115074
Title: Phase I Study of Fluvastatin-Celebrex Association for Optico-chiasmatic Low Grade Gliomas and High Grade Gliomas Localized Outside the Brainstem, Relapsed or Refactory, in Children or Young Adults
Brief Title: Safety of Fluvastatin-Celebrex Association in Low-grade and High Grade Optico-chiasmatic Gliomas
Acronym: FLUVABREX
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Collaborators: Anticancer Fund, Belgium (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FLUVABREX-1208
Record Dates: First submitted 2014-03-26; First posted 2014-04-15 (Estimated); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Glioma
Keywords: Low-grade gliomas; high-grade gliomas; optico-chiasmatic; relapsed; refractory
MeSH Terms: conditions — Glioma; Recurrence | interventions — Fluvastatin; Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fluvastatine Celebrex (Experimental): dose escalation for Fluvastatine
  Interventions: Drug: Fluvastatine; Drug: Celebrex

INTERVENTIONS:
Drug: Fluvastatine — Escalation dose : Level 1: 2mg/kg/day. Level 2: 4mg/kg/day. Level 3: 6mg/kg/day. Level 4: 8mg/kg/day.
  Per os from D1 to D14 of each 28 day cycle.
  Number of Cycles: until progression or unacceptable toxicity develops.
Drug: Celebrex — Dose levels : 100 mg twice a day (< 20 kg), 200 mg twice a day (20-50 kg), 400 mg twice a day (> 50 kg)
  Per os from D1 to D28 of each 28 day cycle.
  Number of Cycles: until progression or unacceptable toxicity develops.
  Other Names: Celecoxib

SUMMARY:
Optico-chiasmatic gliomas have therapeutic feature since surgical resection plays a secondary role. Unlike other sites, many of these tumors are not amenable to complete resection either because of anatomical location, and sometimes they only can be biopsied. A substantial number of children will have recurrences following resection or will experience progression following incomplete tumor removal or biopsy.

Celebrex is a Cox-2 inhibitor with anti-angiogenic and anti-tumor properties, while statins are known to increase the sensitivity of gliomas to anti-tumor agents. Their association could be administered for long periods, in the hope of much reduced risk of toxicities.

This is a national, multicentric, interventional, open-label, non-comparative, and non-randomized phase I study evaluating the maximum tolerated dose of the Fluvastatin in combination with fixed-dose of Celebrex.

This project involves 10 SFCE health centers accustomed to phase I / II studies(Société Française de Lutte contre les Cancers et Leucémies de l'Enfant et de l'Adolescent - French Society for the Fight against Cancer and Leukemia in Children and Adolescents).

DETAILED DESCRIPTION:
Dose escalation scheme only concerns Fluvastatin, and is based on a CRML model (Continual Reassessment Method Lilelihood approach). Dose associated with a probability of DLT closest to 25% will be considered as Recommended Phase 2 Dose (RP2D).

Escalation phase :

Patients will be included by cohort of 2. First patient will be included at the first dose level of Fluvastatin (2mg/kg/day). The second patient will be included only after sufficient time to assess the absence of DLT on first patient. In absence of DLT during the first 28-day cycle, dose escalation will be allowed (4, then 6 and 8 mg/kg/day of Fluvastatin).

The second and all subsequent patients will be treated at the dose level which DLT probability is closest to 25%, without skipping step. Intra-patient dose escalation is not allowed. Treatment will be administered until progression, or unacceptable toxicity for one year. A minimum of 21 patients will be included during the 1st step, including a minimum of 6 patients receiving RP2D.

Expansion phase :

At RP2D, the number of subjects will be increased to reach a total of 14 evaluable patients, in order to better characterize RP2D safety. Patients will be included in the expansion phase according CRML model as well, to confirm the recommended dose.

Probabilities of DLT associated with each dose level will be re-estimated by CRML progressively, without the need to suspend inclusions. Results could modify RP2D retained during 1st step (dose reduction or a dose re-escalation).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed recurrent or progressive primary hypothalamic-chiasmatic low grade glioma, and not warranting a biopsy or surgery
* Histologically confirmed recurrent or progressive primary hypothalamic-chiasmatic high grade glioma, or in complete remission after a new exeresis, excepted brainstem gliomas
* Relapsed or refractory disease after at least 1 line adjuvant treatment including radiation therapy, but not surgery
* Measurable lesions according to RANO criteria for the patients with low grade glioma and for the patients with high grade glioma included in RP2D level (Recommended Phase 2 Dose).
* Non-measurable lesions according to RANO criteria for patients with high grade glioma included in the dose escalation step.
* Age > 6 years and < 21 years old
* Lansky score > 70 or WHO score < 2 (neurological conditions associated with the disease should not be taken into consideration)
* Haematological conditions: ANC > 1000/mm3 and platelets > 75000/mm3
* Creatinine < 1.5 x normal for age or calculated clearance > 70 ml/mn/1.73m2
* Hepatic function: Total bilirubin < 3 N and SGOT and SGPT < 4 N
* Muscle enzymes : CPK < 2 N
* No organ toxicity superior to grade 2 according to NCI-CTCAE v4.0
* No allergy, hypersensibility to one of the compounds of the treatment
* Patients able to swallow capsules
* Life expectancy at least > 6 months for low grade gliomas and > 3 months for high grade gliomas
* Patient affiliated with a health insurance system
* Effective contraception for patients (male and female) with reproductive potential throughout the treatment period
* Written informed consent of patient and/or parents/guardians prior to the study participation

Exclusion Criteria:

* Chemotherapy within 21 days before D1 of experimental treatment. This period may be shortened in case of previous chemotherapy with vincristine (2 weeks), or extended in case of targeted therapies (4 weeks), or treatment by nitrosoureas (6 weeks)
* Radiotherapy within 6 months before D1 of experimental treatment
* Peptic ulcer disease, or gastrointestinal bleeding
* Known hypersensitivity to sulfonamides.
* History of asthma, acute rhinitis, nasal polyps, angioedema, urticaria or other allergic-type reactions induced by acetylsalicylic acid or NSAIDs , including COX-2 inhibitors (cyclo-oxygenase- 2)
* Inflammatory bowel disease.
* Known congestive heart failure (NYHA II- IV)
* Ischemic proven, peripheral and/or history of arterial stroke (including transient ischemic attack)
* Pregnancy or breast feeding woman
* Known allergy to experimental treatment
* Organ toxicity superior to grade 2 according to NCI-CTCAE v4.0
* Active infection
* Pre-existing muscle pathology
* Unsuitable for medical follow-up (geographic, social or mental reasons)

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of Fluvastatine combined to a fixed-dose of Celebrex | 28 days (at the end of the first cycle)
  The MTD is evaluated according to NCI-CTC v4.0 scale, and is defined as follows:
  * grade 3 or 4 neutropenia leading to a delay of therapy superior to 7 days
  * grade 3 or 4 thrombocytopenia requiring transfusions over a period superior to 7 days
  * grade 3 or 4 non-hematologic toxicities, excepted the following events:
    * nausea and vomiting despite appropriate symptomatic treatment,
    * grade 3 fever, and grade 3 liver toxicity but rapidly reversible,
    * grade 3 elevation of creatine phosphokinase (CPK) levels, but rapidly reversible (back <3 X normal within 2 weeks after interruption of treatment)
  * Toxicity leading to dose reduction (<75% dose protocol) will also be considered as a DLT, although the grade of toxicity does not in itself justify this classification

SECONDARY OUTCOMES:
Adverse events | During all the treatment period, for up to 1 year
  Safety is assessed according to NCI-CTC v4.0 scale
Efficacy in terms of overall survival | From date of registration until the date of death from any cause, assessed up to 2 years
  Efficacy is measured according to RANO criteria
Efficacy in terms of progression-free survival | After 3, 6, 9 and 12 months of treatment
  Efficacy is measured according to RANO criteria.
Potential interactions between the two drugs | Pharmacokinetics: 1 blood sample of 1.5 ml is collected during cycle 1 and at day 1 of the second cycle before fluvastatine and celebrex administration.
  The Fluvastatin and Celebrex are dosed on the same sample, then compared with pharmacokinetics data from the literature (when drugs are administered alone). The objective is to explore the interaction between the 2 drugs.
  Pharmacokinetic analysis is performed by liquid chromatography coupled to mass spectrometry (LC/MS), with UV detection.
Best response' s distribution during the treatment | After 3, 6, 9 and 12 months of treatment
  Best response is measured according to RANO criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre LEBLOND, MD, Study Director — Centre Oscar Lambret, Lille, France; Nicolas ANDRE, MD, Study Director — Hôpital pour Enfants de " La Timone " AP-HM, Marseille, France
Locations (8):
- France (8):
  - CHU Angers, Angers
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Hôpital pour enfants La Timone, Marseille
  - Institut Curie, Paris
  - Centre Hospitalier de Strasbourg, Strasbourg
  - Centre Hospitalier de Purpan - Hôpital des Enfants, Toulouse
  - Centre Hospitalier de Nancy, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No